CLINICAL TRIAL: NCT02650453
Title: Ongoing Registry of Deep Venous Reconstructions
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: OP-VE-01
Record Dates: First submitted 2015-12-28; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-12

CONDITIONS: Venous Thrombosis
Keywords: Stent; Angioplasty; Endophlebectomy
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Deep venous reconstruction — PTA & stenting with/without endophlebectomy and/or arteriovenous fistula creation

SUMMARY:
Ongoing registration of deep venous obstructive disease patients treated by means of percutaneous transluminal angioplasty (PTA) and stenting with or without endophlebectomy (surgical desobstruction, also termed endovenectomy) of the common femoral vein and/or arteriovenous fistula creation.

DETAILED DESCRIPTION:
Literature has shown endovenous reconstructions to be safe en effective in treating deep venous obstructive disease. Deep venous obstruction can develop in cases of (iliac) vein compression syndromes (e.g. May-Thurner syndrome) or in cases of post-thrombotic syndrome. In patients with both significant complaints (objectively measured) and venous obstruction objectified on imaging (duplex ultrasonography, magnetic resonance venography, CT-venography) stenting is indicated.

In cases of extensive post-thrombotic damage to the veins of the lower extremity endophlebectomy (surgical desobstruction) of the common femoral vein can be warranted. This operation is generally combined with the creation of an arteriovenous fistula.

Data of patients treated in our tertiary medical centre are entered in a prospective digital database, and continuously updated.

ELIGIBILITY:
Inclusion Criteria:

* Venous obstruction/occlusion in the femoral vein, common femoral vein, external iliac vein, common iliac vein or inferior vena cava

Exclusion Criteria:

* Intolerance to anticoagulant medication
* A life expectancy <1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiënts undergoing deep venous reconstuctive interventions in cases of deep venous obstructive disease; such as (but not limited to) post-thrombotic syndrome and May-Thurner syndrome
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2019-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in patency (primary, assisted primary and secondary) of the treated vein tracts assessed by duplex ultrasonography at regular time intervals. | 2, 6, 12, 23, 52 weeks post-intervention and yearly afterwards
  Patency is defined as the presence of bloodflow as imaged by use of duplex ultrasonography. Patency will be divided in 3 subgroups; primary patency, assisted primary patency and secondary patency.
  Primary patency is defined as presence of bloodflow during follow-up without any interventions undertaken to preserve or reclaim the openness of the treated vein segments.
  Assisted primary patency is defined as the presence of bloodflow during follow-up after use of an intervention to preserve the openness of the treated vein segments.
  Secondary patency is defined as the presence of bloodflow during follow-up after use of an intervention to reclaim the openness of the treated vein segments.

SECONDARY OUTCOMES:
Change in Quality of Life (QoL), assessed by Short form (SF)-36 health survey. | Baseline, 12 and 52 weeks post-intervention, and yearly thereafter.
  The SF-36 is a generic QoL questionnaire.
Change in QoL, assessed by EuroQol 5 Dimensions (EQ-5D) questionnaire. | Baseline, 3 and 12 months post-intervention and yearly afterwards
  The EQ-5D is a generic QoL questionnaire.
Change in QoL, assessed by Venous Insufficiency Epidemiological and Economic Study-quality of life/symptoms scales (VEINES-QoL/sym). | Baseline, 3 and 12 months post-intervention and yearly afterwards
  The VEINES-QoL/sym is a disease-specific QoL questionnaire aimed at venous disease.
Change in Venous Clinical Severity Score (VCSS). | Baseline, 2, 6, 12, 23, 52 weeks post-intervention and yearly afterwards
  The VCSS is a validated scoring system for assessing signs, symptoms and complaints of venous disease.
Change in Villalta scale | Baseline, 2, 6, 12, 23, 52 weeks post-intervention and yearly afterwards
  The Villalta scale is a validated scoring system for assessing signs, symptoms and complaints of the post-thrombotic syndrome.
Venous claudication; number of patients with presence or absence of venous claudication pre-intervention and post-intervention during follow-up. | Baseline, 2, 6, 12, 23, 52 weeks post-intervention and yearly afterwards
  Venous claudication is the pain which develops in patients with obstructive-type venous disease during ambulation and other types of exercise, and which typically subsides when the patient rests in a lying down position or when sitting with elevation of the lower extremity. It is one of the clinically most important symptoms of (obstructive) venous disease. There is currently no validated or internationally accepted scoring system available. We will therefore note the presence of this typical symptom before treatment, and at regular intervals post-intervention (i.e. 2, 6, 12, 23, 52 weeks post-intervention and yearly afterwards).

CONTACTS AND LOCATIONS:
Overall Officials: Cees Wittens, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No